CLINICAL TRIAL: NCT03898960
Title: Post Marketing Study of Patients to Evaluate NIMBUS Revascularization Effectiveness With Challenging Occlusions
Brief Title: Post Marketing Study to Evaluate the NIMBUS Device
Acronym: SPERO
Status: Completed | Type: Observational
Sponsor: Neuravi Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: CNV_2018_01
Record Dates: First submitted 2019-03-29; First posted 2019-04-02 (Actual); Results first posted 2023-11-27 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Cerebral Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Thrombus/Clot
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mechanical Thrombectomy: NIMBUS Device
  Interventions: Device: NIMBUS Device

INTERVENTIONS:
Device: NIMBUS Device — NIMBUS Geometric Clot Extractor

SUMMARY:
A post-market study evaluating the NIMBUS Device in acute ischemic stroke patients with confirmed intracranial large vessel occlusion.

DETAILED DESCRIPTION:
The objective of this study is to assess the efficacy of the NIMBUS Device. The study will also report on clot characteristics and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* The subject or the subject's legally authorized representative has signed and dated an Informed Consent Form.
* Patient has had one or two passes of another mechanical thrombectomy device without achieving mTICI 2b or better and continues to have angiographic confirmation of a Large Vessel Occlusion (LVO) in the same vessel.
* mRS 0-1 prior to this stroke.
* NIMBUS is used on the second or third overall pass to attempt revascularization.

Exclusion Criteria:

* Currently participating in an investigational (drug, device, etc.) clinical trial that may confound study endpoints. Patients in observational, natural history, and/or epidemiological studies not involving intervention are eligible.
* Confirmation of positive pregnancy test according to site specific standard of care (e.g. test, verbal communication).
* All patients with severe hypertension on presentation (SBP > 220 mmHg and/or DBP > 120 mm Hg). All patients, in whom intravenous therapy with blood pressure medications is indicated, with hypertension that remains severe and sustained despite intravenous antihypertensive therapy (SBP >185 mmHg and/ or DBP >110 mmHg).
* Known cerebral vasculitis.
* Known cancer with life expectancy less than 12 months.
* Stenosis, or any occlusion, in a proximal vessel that requires treatment or prevents access to the site of occlusion.
* Intracranial stenosis that prevents access to the site of occlusion.
* Computed tomography (CT) or Magnetic Resonance Imaging (MRI) evidence of recent/ fresh hemorrhage on presentation.
* Baseline computed tomography (CT) or MRI showing mass effect or intracranial tumor (except small meningioma).
* Evidence of dissection in the extra or intracranial cerebral arteries.
* Occlusions in multiple vascular territories (e.g., bilateral anterior circulation, or anterior/posterior circulation).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute Ischemic Stroke patients with confirmed intracranial Large Vessel Occlusion.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2019-10-30 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-04-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: René van den Berg, MD, PhD, Principal Investigator — Amsterdam UMC
Locations (2):
- UKE Hamburg, Hamburg, Germany
- Karolinska Institute, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu.
URL: http://yoda.yale.edu

REFERENCES:
- [Derived] van den Berg R, Ribo M, Arnberg Sandor F, Estrade L, Thornton J, Tomasello A, Gontu V, Hernandez D, Karam A, Bricout N, Buhk JH, Clarencon F, Desal H, Januel AC, Nouri N, Wiesmann M, Doyle K, Liebeskind DS, McManus C, Mirza M, Andersson T, Brouwer P. Post-marketing study of patients to evaluate NIMBUS revascularization effectiveness with challenging occlusions (SPERO): study results. J Neurointerv Surg. 2026 Jan 6:jnis-2025-023811. doi: 10.1136/jnis-2025-023811. Online ahead of print. PMID 41494867

RESULTS

PARTICIPANT FLOW:
Groups:
- Mechanical Thrombectomy: NIMBUS Device: Participants with acute ischemic stroke who had post one or two unsuccessful passes of another mechanical thrombectomy therapy and did not achieve modified thrombolysis in cerebrovascular infarction (mTICI) 2b or better, were treated with NIMBUS device.
Period: Overall Study
Arm/Group | Mechanical Thrombectomy: NIMBUS Device
Started | 54
Completed | 44
Not Completed | 10
Not completed — Death | 10

BASELINE CHARACTERISTICS:
Arm/Group | Mechanical Thrombectomy: NIMBUS Device
Number analyzed (Participants) | 54
Age, Continuous [Mean (Standard Deviation); unit: Years] | 71.9 (14.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 22
  More than one race | 0
  Unknown or Not Reported | 31

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Successful Revascularization With NIMBUS Device
Description: Successful revascularization was defined as achieving an modified thrombolysis in cerebrovascular infarction (mTICI) score of 2b or greater as determined by an Independent Core Laboratory. The expanded treatment in cerebral infarction (eTICI) score was a modified from the mTICI scale. eTICI was a 6-point grading system for determining the response of thrombolytic therapy for ischemic stroke: 0=No reperfusion; 0 percent (%) filling of the downstream territory; 1=Thrombus reduction without any reperfusion of distal arteries; 2a=Reperfusion in less than half (1-49%) of the territory; 2b=2b50 (reperfusion in [50-66%] of downstream territory) and 2b67 (reperfusion in (67-89%) of downstream territory); 2c=Reperfusion in [90-99%] of downstream territory; 3=Complete and 100% reperfusion.
Time Frame: Day 1
Population: The modified intent-to-treat (mITT) analysis set consisted of all participants who were enrolled into the study, and who had attempted at least one pass with the NIMBUS device (which included deployment and retrieval with the NIMBUS device). Here 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Mechanical Thrombectomy: NIMBUS Device
Number analyzed (Participants) | 51
Percentage of participants | 68.6 [54.1 to 80.9]

2. Secondary Outcome: Percentage of Participants With Successful Procedural Revascularization
Description: Successful procedural revascularization was defined as achieving an mTICI score of 2b or greater at the end of procedure as determined by an Independent Core Laboratory. The eTICI score was a modified from the mTICI scale. eTICI was a 6-point grading system for determining the response of thrombolytic therapy for ischemic stroke: 0=No reperfusion; 0% filling of the downstream territory; 1=Thrombus reduction without any reperfusion of distal arteries; 2a=Reperfusion in less than half (1-49%) of the territory; 2b=2b50 (reperfusion in [50-66%] of downstream territory) and 2b67 (reperfusion in [67-89%] of downstream territory); 2c=Reperfusion in [90-99%] of downstream territory; 3=Complete and 100% reperfusion.
Time Frame: Day 1
Population: The mITT analysis set consisted of all participants who were enrolled into the study, and who had attempted at least one pass with the NIMBUS device (which included deployment and retrieval with the NIMBUS device). Here 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Mechanical Thrombectomy: NIMBUS Device
Number analyzed (Participants) | 53
Percentage of participants | 79.2 [65.9 to 89.2]

3. Secondary Outcome: Percentage of Participants With Excellent Procedural Revascularization
Description: Excellent procedural revascularization was defined as achieving an mTICI score of 2c or greater at the end of procedure as determined by an Independent Core Laboratory. The eTICI score was a modified from the mTICI scale. eTICI was a 6-point grading system for determining the response of thrombolytic therapy for ischemic stroke: 0=No reperfusion; 0% filling of the downstream territory; 1=Thrombus reduction without any reperfusion of distal arteries; 2a=Reperfusion in less than half (1-49%) of the territory; 2b=2b50 (reperfusion in [50-66%] of downstream territory) and 2b67 (reperfusion in [67-89%] of downstream territory); 2c=Reperfusion in (90-99%) of downstream territory; 3=Complete and 100% reperfusion.
Time Frame: Day 1
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Mechanical Thrombectomy: NIMBUS Device
Number analyzed (Participants) | 53
Percentage of participants | 37.7 [24.8 to 52.1]

4. Secondary Outcome: Percentage of Participants With First Pass Revascularization Using NIMBUS Device
Description: First Pass revascularization was defined as achieving an mTICI score of 2b or greater after the first use of NIMBUS device as determined by an Independent Core Laboratory. The eTICI score was a modified from the mTICI scale. eTICI was a 6-point grading system for determining the response of thrombolytic therapy for ischemic stroke: 0=No reperfusion; 0% filling of the downstream territory; 1=Thrombus reduction without any reperfusion of distal arteries; 2a=Reperfusion in less than half (1-49%) of the territory; 2b=2b50 (reperfusion in [50-66%] of downstream territory) and 2b67 (reperfusion in [67-89%] of downstream territory); 2c=Reperfusion in (90-99%) of downstream territory; 3=Complete and 100% reperfusion.
Time Frame: Day 1
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Mechanical Thrombectomy: NIMBUS Device
Number analyzed (Participants) | 51
Percentage of participants | 52.9 [38.5 to 67.1]

5. Secondary Outcome: Percentage of Participants With Embolization to a New Territory (ENT)
Description: Percentage of participants with ENT was reported.
Time Frame: Day 1
Population: The mITT analysis set consisted of all participants who were enrolled into the study, and who had attempted at least one pass with the NIMBUS device (which included deployment and retrieval with the NIMBUS device).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Mechanical Thrombectomy: NIMBUS Device
Number analyzed (Participants) | 54
Percentage of participants | 0 [0.0 to 6.6]

6. Secondary Outcome: Percentage of Participants With Symptomatic Intracerebral Hemorrhage (sICH) According to the Heidelberg Bleeding Classification (HBC)
Description: Percentage of participants with sICH according to the HBC was reported. sICH was defined as new intracranial hemorrhage detected by brain imaging associated with any of the item: greater than or equal to (>=) 4 points total National Institute of Health Stroke Scale (NIHSS) at the time of diagnosis compared to immediately before worsening; >=2 point in one NIHSS category. The rationale for this was to capture new hemorrhages that produce new neurological symptoms, making them clearly symptomatic but not causing worsening in the original stroke territory; leading to intubation/hemicraniectomy/external ventricular drain (EVD) placement or other major medical/surgical intervention; absence of alternative explanation for deterioration.
Time Frame: Day 1
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Mechanical Thrombectomy: NIMBUS Device
Number analyzed (Participants) | 54
Percentage of participants | 3.7 [0.5 to 12.7]

7. Secondary Outcome: Number of Participants With All-Cause Mortality
Description: Number of participants with all-cause mortality at 90 days post-procedure on Day 0 was reported. All-cause mortality included all deaths of participants due to any cause.
Time Frame: Up to Day 90
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Mechanical Thrombectomy: NIMBUS Device
Number analyzed (Participants) | 54
Participants | 10

8. Secondary Outcome: Percentage of Participants With Modified Rankin Scale (mRS) Score of Less Than or Equal to (<=) 2
Description: Percentage of participants with mRS score of <=2 was reported. The mRS was a 7-point scale that ranged from 0 to 6 where 0=no symptoms at all; 1=no significant disability despite symptoms; 2=slight disability; 3=moderate disability; 4=moderately severe disability; 5=severe disability; 6=death.
Time Frame: Up to Day 90
Population: The mRS analysis set consisted of all mITT participants who met study criteria as MRI criterion: volume of diffusion restriction visually assessed <=50 milliliter(mL), computed tomography(CT) criterion: ASPECTS 6 to 10 on baseline CT, computed tomography angiography(CTA)-source images or volume of significantly lowered cerebral blood volume(CBV) <=50 mL; NIHSS >=8 and less than (<)30; participants treated within 6 hours of onset of stroke symptoms (start of treatment defined as groin puncture).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Mechanical Thrombectomy: NIMBUS Device
Number analyzed (Participants) | 15
Percentage of participants | 46.7 [21.3 to 73.4]

ADVERSE EVENTS:
Time Frame: Up to Day 90
Description: Safety set included all participants who were enrolled into the study, and who had attempted at least one pass with the NIMBUS device (which included deployment and retrieval with the NIMBUS device).
Arm/Group | Mechanical Thrombectomy: NIMBUS Device
All-Cause Mortality (participants affected / at risk) | 10/54
Serious Adverse Events (participants affected / at risk) | 21/54
Other Adverse Events (participants affected / at risk) | 6/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mechanical Thrombectomy: NIMBUS Device (N=54)
Stroke in evolution (Nervous system disorders) | 4 (4)
Hemorrhagic transformation stroke (Nervous system disorders) | 3 (3)
Brain oedema (Nervous system disorders) | 1 (1)
Cerebral hemorrhage (Nervous system disorders) | 1 (1)
Ischemic stroke (Nervous system disorders) | 1 (1)
Subarachnoid hemorrhage (Nervous system disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bacteriuria (Infections and infestations) | 1 (1)
Bronchitis hemophilus (Infections and infestations) | 1 (1)
Endocarditis (Infections and infestations) | 1 (1)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mechanical Thrombectomy: NIMBUS Device (N=54)
Stroke in evolution (Nervous system disorders) | 1 (1)
Hemianopia (Nervous system disorders) | 1 (1)
Partial seizures (Nervous system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 1 (1)
Vascular access site pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Draft abstracts, manuscripts, and materials for presentation at scientific meetings must be sent to the sponsor at least 60 working days prior to abstract or other relevant submission deadlines. Authorship of publications resulting from this study was based on generally accepted criteria for major medical journals.

DOCUMENTS (2):
  • Study Protocol (2020-07-23): https://cdn.clinicaltrials.gov/large-docs/60/NCT03898960/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-25): https://cdn.clinicaltrials.gov/large-docs/60/NCT03898960/SAP_001.pdf